CLINICAL TRIAL: NCT02881983
Title: Study of Mechanisms of Emotion Regulation in Short- and Long-term Alcohol-abstinent Patients
Brief Title: Study of Mechanisms of Emotion Regulation in Alcohol-abstinent Patients
Acronym: REAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_31; 2014-A00105-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; emotion processing; abstinence; sympathetic system; parasympathetic system
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- STA group: Short-term alcohol abstinent patients (after 1 month of withdrawal)
  Interventions: Other: the presentation of pictures (static stimuli) or videos (dynamic stimuli)
- LTA group: Long-term alcohol abstinent patients (at least 6 months of abstinence)
  Interventions: Other: the presentation of pictures (static stimuli) or videos (dynamic stimuli)
- Control group: Healthy subjects
  Interventions: Other: the presentation of pictures (static stimuli) or videos (dynamic stimuli)

INTERVENTIONS:
Other: the presentation of pictures (static stimuli) or videos (dynamic stimuli)

SUMMARY:
Background:

Difficulties in assigning and identifying emotional states, or to regulate the emotional costs are recognized as one of the major factors of relapse. This study aimed to evaluate the emotion regulation processes, in short term (STA, after 1month of withdrawal) and long-term alcohol abstinent individuals (LTA, at least six months of abstinence), compared to healthy control participants (C) in a positive and negative emotion induction protocol.

Main aim:

Evaluating the emotional regulation deficits assessed with physiological indicators (heart rate variability, electrodermal response, pupil diameter) and clinically in presentations of visual stimuli to emotional value (positive, negative, neutral) in alcohol use disorder's (AUD) patients with short and long term abstinent compared to a control group of healthy subjects. The investigators are particularly interested in the evolution of heart rate variability considered as a good marker of vulnerability to AUD.

Secondary objectives:

Studying the relationships between physiological measures and clinical variables such as behavioral indicators and self-reported assessment of cognitive and emotional skills among the three groups (STA, LTA and C).

DETAILED DESCRIPTION:
The recording was performed for all participants during presentation of high emotional inducing stimuli presenting human interactions (pictures and video sequences). For each participant physiological responses (pupil diameter, heart rate, and skin conductance) were recorded before, during and after induction.

Participants were asked to evaluate the intensity and the valence of emotional stimuli.

In addition, a neurological evaluation, a clinical and cognitive assessment were performed.

Neurological, clinical and cognitive evaluation - Each participant had a clinical structured interview, a neurological evaluation, self-administered assessment (Hospital Anxiety & Depression Scale, Emotional Skills Profile, Obsessive Compulsive Drinking Scale, and cognitive assessment (Montreal Cognitive Assessment).

Physiological assessment - The recording was performed for all participants during the presentation of pictures (static stimuli) or videos (dynamic stimuli) selected according to their high emotional intensity (positive, neutral and negative valence), representing human interactions. For each participant heart rate, electrodermal activity, and pupil diameter were recorded during three experimental conditions: rest, induction (presentation of stimuli) and after induction (recovery). Participants were asked to evaluate the intensity and valence of the pictures and videos using the Self-Assessment Manikin.

ELIGIBILITY:
Inclusion Criteria:

For STA and LTA groups :

* a diagnosis of severe alcohol use disorder (DSM5 criteria, 2013 confirmed by an addictonologist and a psychologist),
* successful completion of withdrawal,
* an intended treatment length of at least 1 month (for the STA group) or at least 6 months (for the LTA group).

For Control participants (C) :

- social drinkers, and were recruited from the general population (e.g. at the university).

Exclusion Criteria:

* with delusional psychiatric disorders (and/or medication for psychiatric disorders (excepted anxiolytics),
* neurological or cardiological disorders,
* taking medication that may act on heart rate or alter the regulation of body temperature or cognitive functions,
* with active co-dependence (except for tobacco)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Short term alcohol abstinent patients (STA, after 1month of withdrawal)
  * Long-term alcohol abstinent individuals (at least six months of abstinence)
  * Healthy control participants (C)
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 3 years
  High measuring heart rate

SECONDARY OUTCOMES:
Electrodermal response | 3 years
  skin conductance
pupil diameter | 3 years
  pupil diameter
HAD score | 3 years
  Score at the Hospital Anxiety & Depression Scale
MocA assessment | 3 years
  Montréal cognitive Assessement score

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - CSAPA, Lille
  - CHRU Lille, Fontan2, Lille

IPD SHARING:
Plan to Share IPD: No